CLINICAL TRIAL: NCT04444895
Title: An Open-Label Study to Evaluate the Long-Term Safety and Efficacy of Lanadelumab for Prevention Against Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH)
Brief Title: A Study of Long-Term Safety and Efficacy of Lanadelumab for Prevention of Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-743-3001; 2019-004823-20 (EudraCT Number); jRCT2051220001 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Angioedema
MeSH Terms: conditions — Angioedema | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lanadelumab 300 mg Every 2 Weeks (Experimental): Participants received 300 milligrams (mg) lanadelumab subcutaneous (SC) injection, every 2 weeks (Q2W) for up to 26 weeks with an option to switch to lanadelumab 300 mg every 4 weeks (Q4W) if attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor.
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Lanadelumab SC injection
  Other Names: DX-2930; SHP643; TAK-743

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of repeated subcutaneous (SC) administration of lanadelumab in adolescents and adults with non-histaminergic angioedema with normal C1-inhibitor who completed study SHP643-303 (NCT04206605).

DETAILED DESCRIPTION:
This study consists of 26-week treatment period (Day 0 to Day 182) and a 2-week follow-up period. Participants who completed the double-blind treatment period at Day 182 of Study SHP643-303 (NCT04206605) will enroll into this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 12 years of age and older diagnosed with non-histaminergic normal C1-INH angioedema at the time of enrollment into the antecedent Study SHP643-303 (NCT04206605).
* Participants must have completed the treatment period (through Visit 26/Day 182) of Study SHP643-303 (NCT04206605) without reporting a clinically significant TEAE that would preclude subsequent exposure to lanadelumab.
* Agree to adhere to the protocol-defined schedule of treatments, assessments, and procedures.
* Males, or non-pregnant, non-lactating females who are of child-bearing potential and who agree to be abstinent or agree to comply with the applicable contraceptive requirements of this protocol for the duration of the study; or females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months.
* The participant (or the participant's parent/legal guardian, if applicable) has provided written informed consent approved by the institutional review board/research ethics board/ethics committee (IRB/REB/EC) at any time prior to study start. If the participant is a minor (i.e. lesser then (<) 18 years of age), have a parent/legal guardian who is informed of the nature of the study provide written informed consent (i.e. permission) for the minor to participate in the study before any study-specific procedures are performed. Assent will be obtained from minor participants.

Exclusion Criteria:

* Discontinued from Study SHP643-303 (NCT04206605) after enrollment but before Visit 26 for any reason.
* Presence of important safety concerns identified in Study SHP643-303 (NCT04206605) that would preclude participation in this study.
* Dosing with an investigational product (IP, not including IP defined in antecedent Study SHP643-303 [NCT04206605]) or exposure to an investigational device within 4 weeks prior to Day 0.
* Participants has a known hypersensitivity to the investigational product or its components.
* Have any condition (surgical or medical) that, in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude the successful conduct of the study, or interfere with interpretation of the results (e.g. significant pre-existing illness or other major comorbidities that the investigator considers may confound the interpretation of study results).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas
Locations (35):
- United States (15):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - UCSD Angioedema Center, San Diego, California
  - Allergy and Asthma Clinical Research Inc, Walnut Creek, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Kanarek Allergy, Asthma and Immunology, Overland Park, Kansas
  - Institute for Asthma & Allergy, P.C., Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington
- Canada (2):
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec
- Hôpital Saint-Antoine, Paris, France
- Germany (2):
  - Klinikum rechts der Isar der TU, Munich, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet pt, Frankfurt am Main, Hesse
- Semmelweis Egyetem, Budapest, Hungary
- Italy (4):
  - A.O. Ospedali riuniti Villa Sofia - Cervello,, Palermo, Palermo Palermo
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
- Japan (3):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kobe University Hospital, Kobe, Hyōgo
  - Clover Hospital, Fujisawa-shi, Kanagawa
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Poland (2):
  - NZOZ Homeo Medicus, Poradnia Alergologiczna, Bialystok
  - "ALL-MED" Specjalistyczna Opieka Medyczna Filia, Wroclaw
- Spain (2):
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Riedl MA, Staubach P, Farkas H, Zanichelli A, Ren H, Nurse C, Andresen I, Juethner S, Yu M, Zhang J. Lanadelumab for prevention of attacks of non-histaminergic normal C1 inhibitor angioedema: results from the randomized, double-blind CASPIAN Study and CASPIAN open-label extension. Front Immunol. 2025 May 21;16:1502325. doi: 10.3389/fimmu.2025.1502325. eCollection 2025. PMID 40469312
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b600d4db2bf003ab48cf1?idFilter=%5B%22TAK-743-3001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 73 participants took part in the study at 34 investigative sites in Canada, France, Germany, Hungary, Italy, Japan, Netherlands, Poland, Spain, and the United States from 05 February 2021 to 05 May 2023.
Pre-assignment Details: Participants with a diagnosis of non-histaminergic angioedema rolled over from the study SHP643-303 (NCT04206605) to receive lanadelumab 300 mg every 2 weeks (Q2W) of whom 2 participants switched to lanadelumab 300 mg at a reduced frequency of every 4 weeks (Q4W) for some time during the study.
Groups:
- Lanadelumab 300 mg Q2W: Participants received 300 milligrams (mg) lanadelumab subcutaneous (SC) injection, every 2 weeks (Q2W) for up to 26 weeks with an option to switch to lanadelumab 300 mg every 4 weeks (Q4W) if attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor.
Period: Overall Study
Arm/Group | Lanadelumab 300 mg Q2W
Started | 73
Reduced-dose Safety AnalysisSet(RD-SFAS) (The RD-SFAS Set was a subset of the Safety Analysis Set (SFAS) and included participants who switched from lanadelumab 300 mg Q2W to a lanadelumab 300 mg Q4W dosing regimen as recorded on the Dose Frequency Modification electronic case report form.) | 2
Completed | 64
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab).
Groups:
- Lanadelumab 300 mg Q2W: Participants received 300 mg lanadelumab SC injection, Q2W for up to 26 weeks with an option to switch to lanadelumab 300 mg Q4W if attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor.
Arm/Group | Lanadelumab 300 mg Q2W
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 64
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5
  France | 1
  Germany | 3
  Hungary | 2
  Italy | 7
  Japan | 4
  Netherlands | 3
  Poland | 6
  Spain | 3
  United States | 39
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number of participants analyzed is the number of participants with data available for weight at the Baseline.
  kilograms (kg)
    number analyzed (Participants) | 72
    (all) | 81.52 (23.129)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 166.75 (8.938)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI= weight(kg) / height(meter)^2 Population: Number of participants analyzed is the number of participants with data available for BMI at the Baseline.
  kilogram per square meter (kg/m^2)
    number analyzed (Participants) | 72
    (all) | 29.23 (7.972)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs) During Treatment Period
Description: TEAE: Any event emerging or manifesting at or after initiation of treatment with investigational product (IP) or medicinal product or any existing event that worsens in either intensity or frequency following exposure to IP or medicinal product including clinically meaningful findings in laboratory safety tests, vital signs, weight, and electrocardiogram (ECG) findings. SAE: Any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to IP or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event. AESI included hypersensitivity reactions, events of disordered coagulation such as bleeding AESI, hypercoagulable AESI. TEAEs were classified and reported as angioedema attack and non-angioedema attack adverse events in this outcome measure.
Time Frame: From Day 0 up to Day 182
Population: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab). The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Measure: Count of Participants; unit: Participants
Groups:
- Lanadelumab 300 mg Q4W: Participants who received 300 mg lanadelumab, SC injection, Q4W as attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor at any point during the 26-week treatment period were included in this group.
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
Participants
  Any TEAEs: Non-Angioedema Attack | 55 | 1
  Any TEAEs: Angioedema Attack | 61 | 1
  AESI: Non-Angioedema Attack | 1 | 0
  AESI: Angioedema Attack | 0 | 0
  Any SAEs: Non-Angioedema Attack | 5 | 1
  Any SAEs: Angioedema Attack | 3 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs) During Follow-up
Description: as for outcome 1
Time Frame: From Day 183 up to Day 196
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
Participants
  Any TEAEs: Non-Angioedema Attack | 4 | 0
  Any TEAEs: Angioedema Attack | 19 | 0
  AESI: Non-Angioedema Attack | 0 | 0
  AESI: Angioedema Attack | 0 | 0
  Any SAEs: Non-Angioedema Attack | 0 | 0
  Any SAEs: Angioedema Attack | 0 | 0

3. Secondary Outcome: Number of Investigator-Confirmed Angioedema Attacks During the Treatment Period of Day 0 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of investigator-confirmed angioedema attacks during the treatment period of Day 0 through Day 182 was assessed.
Time Frame: From Day 0 up to Day 182
Population: as for outcome 1
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
angioedema attacks | 595 | 2

4. Secondary Outcome: Number of Moderate or Severe Angioedema Attacks During the Treatment Period of Day 0 Through Day 182
Description: The overall severity of angioedema attack was determined by the site using following definitions: mild (transient or mild discomfort), moderate (mild to moderate limitation in activity), severe (marked limitation in activity). Number of moderate or severe angioedema attacks during the treatment period of Day 0 through Day 182 was assessed.
Time Frame: From Day 0 up to Day 182
Population: as for outcome 1
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
angioedema attacks | 391 | 2

5. Secondary Outcome: Number of High-Morbidity Angioedema Attacks During the Treatment Period of Day 0 Through Day 182
Description: A high-morbidity angioedema attack was defined as any attack that has at least one of the following characteristics: severe, results in hospitalization (except hospitalization for observation <24 hours), hemodynamically significant (systolic blood pressure (BP) <90 millimetres of mercury (mmHg), requires intravenous hydration, or associated with syncope or near-syncope) or laryngeal.
Time Frame: From Day 0 up to Day 182
Population: as for outcome 1
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
angioedema attacks | 232 | 1

6. Secondary Outcome: Pharmacokinetic (PK) Plasma Concentrations of Lanadelumab
Description: The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Time Frame: Predose on Days 0, 84, and 140 and postdose on Day 182
Population: The Pharmacokinetic (PK) Set included all participants in the SFAS who had at least 1 evaluable postdose PK concentration value. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 68 | 2
nanograms per milliliter (ng/mL)
  Day 0 | 14419.068 (13208.1952) | NA (NA) — The data were not estimable as the values were below the lower limit of quantification.
  Day 84: number analyzed (Participants) | 64 | 1
  Day 84 | 17021.002 (10116.5279) | 7047.860 (NA) — The standard deviation was not estimable for a single participant.
  Day 140: number analyzed (Participants) | 65 | 1
  Day 140 | 21138.057 (12076.9186) | 4944.010 (NA) — The standard deviation was not estimable for a single participant.
  Day 182: number analyzed (Participants) | 68 | 1
  Day 182 | 18799.596 (12054.1105) | 14573.340 (NA) — The standard deviation was not estimable for a single participant.

7. Secondary Outcome: Plasma Kallikrein (pKal) Activity
Description: Plasma kallikrein activity was measured by biomarker cleaved high molecular weight kininogen (cHMWK) with factor XIIa activation level to assess the pharmacodynamics of lanadelumab. The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Time Frame: Predose on Days 0, 84, and 140 and postdose on Day 182
Population: The Pharmacodynamic (PD) Set included all participants in the SFAS who had at least 1 evaluable postdose PD concentration value. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: percentage of cHMWK
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 67 | 2
percentage of cHMWK
  Day 0 | 15.306 (15.2413) | NA (NA) — The data were not estimable as the values were below the lower limit of quantification.
  Day 84: number analyzed (Participants) | 63 | 1
  Day 84 | 17.586 (9.2437) | 21.600 (NA) — The standard deviation was not estimable for a single participant.
  Day 140: number analyzed (Participants) | 64 | 1
  Day 140 | 17.238 (9.1590) | 44.700 (NA) — The standard deviation was not estimable for a single participant.
  Day 182: number analyzed (Participants) | 67 | 1
  Day 182 | 15.515 (9.2074) | 37.100 (NA) — The standard deviation was not estimable for a single participant.

8. Secondary Outcome: Number of Participants With Neutralizing Antidrug Antibodies (ADA) in Plasma
Description: Number of participants with positive ADA including evaluation of neutralizing antibodies in plasma was assessed. As pre-specified in the statistical analysis plan (SAP), data for this outcome measure was collected and analyzed as a single group irrespective of dosing regimen.
Time Frame: Predose on Days 0, 84, and 140 and postdose on Day 182
Population: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab). Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg Q2W
Number analyzed (Participants) | 72
Participants
  Day 0 | 2
  Day 84: number analyzed (Participants) | 65
  Day 84 | 2
  Day 140: number analyzed (Participants) | 66
  Day 140 | 3
  Day 182: number analyzed (Participants) | 69
  Day 182 | 4

9. Secondary Outcome: Change From Baseline in Total Angioedema Quality of Life (AE-QoL) Questionnaire Total Score at End of Treatment Period
Description: The AE-QoL questionnaire is self-administered validated instrument to assess health related (HR)QoL among participants with recurrent angioedema(including hereditary angioedema[HAE]). It consists of 17 disease-specific QOL items, to produce total AE-QoL score & 4 domain scores(functioning,fatigue/mood,fear/shame,nutrition) each of 17 items had 5-point response scale ranging from 1(Never) to 5(Very Often). It was scored according to developers' guidelines to produce 4 domain scores yielding total score. The raw total score(mean of all item scores) was rescaled using linear transformations into final percentage scores ranging 0-100, based on maximum possible score, where higher score, greater QoL impairment. Negative change from Baseline indicates better QoL. Baseline: Last non-missing value prior to first exposure to study drug(based on date or date/time). As pre-specified in SAP, data for this outcome measure was collected and analyzed as single group irrespective of dosing regimen.
Time Frame: Baseline (Day 0) up to end of treatment period (Day 182)
Population: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab). Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lanadelumab 300 mg Q2W
Number analyzed (Participants) | 66
score on a scale | -12.73 (20.696)

10. Secondary Outcome: Number of Participants With Any Pause During Injection
Description: An injection report was completed by the participant (or parent/caregiver) following each dose administration of lanadelumab injection used during the treatment period and any kind of pause during injection was captured. Categories with at least one participant with event are reported.
Time Frame: Days 0, 14, 28, 42, 56, 70, 84, 98, 112, 126, 140, 154, and 168
Population: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab). Number analyzed is the number of participants with data available for analysis at the specified time point. The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 73 | 2
Participants
  Day 0: number analyzed (Participants) | 72 | 1
  Day 0 | 3 | 0
  Day 14: number analyzed (Participants) | 72 | 0
  Day 14 | 5 | 0
  Day 28: number analyzed (Participants) | 70 | 1
  Day 28 | 5 | 0
  Day 42: number analyzed (Participants) | 70 | 0
  Day 42 | 3 | 0
  Day 56: number analyzed (Participants) | 70 | 1
  Day 56 | 3 | 0
  Day 70: number analyzed (Participants) | 70 | 0
  Day 70 | 4 | 0
  Day 84: number analyzed (Participants) | 66 | 2
  Day 84 | 4 | 0
  Day 98: number analyzed (Participants) | 66 | 0
  Day 98 | 1 | 0
  Day 112: number analyzed (Participants) | 67 | 1
  Day 112 | 2 | 1
  Day 126: number analyzed (Participants) | 67 | 0
  Day 126 | 2 | 0
  Day 140: number analyzed (Participants) | 63 | 1
  Day 140 | 3 | 0
  Day 154: number analyzed (Participants) | 64 | 0
  Day 154 | 2 | 0
  Day 168: number analyzed (Participants) | 63 | 1
  Day 168 | 1 | 0

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs) in Participants Who Switched Dosing Regimen
Description: as for outcome 1
Time Frame: From Day 0 up to Day 196
Population: The RD-SFAS Set was a subset of the SFAS Set and included participants who switched from lanadelumab 300 mg Q2W to a lanadelumab 300 mg Q4W dosing regimen as recorded on the Dose Frequency Modification electronic case report form. The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Measure: Count of Participants; unit: Participants
Groups:
- Lanadelumab 300 mg Q2W: Participants who received 300 mg lanadelumab SC injection, Q2W, and switched to the Q4W regimen as attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor at any point during the 26-week treatment period were included in this group.
- Lanadelumab 300 mg Q4W: Participants who received 300 mg lanadelumab SC injection, Q4W as attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor at any point during the 26-week treatment period were included in this group.
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 2 | 2
Participants
  Any TEAEs: Non-Angioedema Attack | 2 | 1
  Any TEAEs: Angioedema Attack | 0 | 1
  AESI: Non-Angioedema Attack | 0 | 0
  AESI: Angioedema Attack | 0 | 0
  Any SAEs: Non-Angioedema Attack | 0 | 1
  Any SAEs: Angioedema Attack | 0 | 0

12. Secondary Outcome: Number of Investigator-Confirmed Angioedema Attacks During the Treatment Period of Day 0 Through Day 182 in Participants Who Switched Dosing Regimen
Description: as for outcome 3
Time Frame: From Day 0 up to Day 182
Population: as for outcome 11
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 2 | 2
angioedema attacks | 0 | 2

13. Secondary Outcome: Number of Moderate or Severe Angioedema Attacks During the Treatment Period of Day 0 Through Day 182 in Participants Who Switched Dosing Regimen
Description: as for outcome 4
Time Frame: From Day 0 up to Day 182
Population: as for outcome 11
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 2 | 2
angioedema attacks | 0 | 2

14. Secondary Outcome: Number of High-Morbidity Angioedema Attacks During the Treatment Period of Day 0 Through Day 182 in Participants Who Switched Dosing Regimen
Description: A high-morbidity angioedema attack was defined as any attack that has at least one of the following characteristics: severe, results in hospitalization (except hospitalization for observation <24 hours), hemodynamically significant (systolic BP <90 mmHg, requires intravenous hydration, or associated with syncope or near-syncope) or laryngeal.
Time Frame: From Day 0 up to Day 182
Population: as for outcome 11
Measure: Number; unit: angioedema attacks
Arm/Group | Lanadelumab 300 mg Q2W | Lanadelumab 300 mg Q4W
Number analyzed (Participants) | 2 | 2
angioedema attacks | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first study drug administration up to follow-up (Day 196)
Description: The SFAS included all participants who received any study drug after entering this study (i.e., any exposure to open-label lanadelumab). The data was partitioned by dosing regimen and reported accordingly to appropriately attribute to each dosing regimen.
Groups:
- Lanadelumab 300 mg Every 2 Weeks: Participants received 300 mg lanadelumab SC injection, Q2W for up to 26 weeks with an option to switch to lanadelumab 300 mg Q4W if attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor.
- Lanadelumab 300 mg Every 4 Weeks: Participants who received 300 mg lanadelumab, SC injection, Q4W as attacks were well-controlled based on the investigator's discretion and consultation with the sponsor's medical monitor at any point during the 26-week treatment period were included in this group.
Arm/Group | Lanadelumab 300 mg Every 2 Weeks | Lanadelumab 300 mg Every 4 Weeks
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/2
Serious Adverse Events (participants affected / at risk) | 7/73 | 1/2
Other Adverse Events (participants affected / at risk) | 65/73 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab 300 mg Every 2 Weeks (N=73) | Lanadelumab 300 mg Every 4 Weeks (N=2)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0
Arthritis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab 300 mg Every 2 Weeks (N=73) | Lanadelumab 300 mg Every 4 Weeks (N=2)
Angioedema (Skin and subcutaneous tissue disorders) | 61 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0
COVID-19 (Infections and infestations) | 17 | 0
Eye swelling (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Headache (Nervous system disorders) | 10 | 1
Injection site pain (General disorders) | 8 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 0
Malaise (General disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04444895/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04444895/SAP_001.pdf